CLINICAL TRIAL: NCT05300763
Title: Clinical Performance of Senofilcon A Investigational Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-6481
Record Dates: First submitted 2022-03-18; First posted 2022-03-29 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TEST LENS (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomly assigned the TEST Lens for the duration of the study.
  Interventions: Device: senofilcon A prototype
- CONTROL LENS (Experimental): Eligible subjects who are habitual soft contact lens wearers will be randomly assigned the CONTROL Lens for the duration of the study.
  Interventions: Device: Dailies Total 1

INTERVENTIONS:
Device: senofilcon A prototype — Test
  Arms: TEST LENS
Device: Dailies Total 1 — Control
  Arms: CONTROL LENS

SUMMARY:
This study is a controlled, randomized, subject-masked, 2-arm parallel, 2-week dispensing, bilateral evaluation where the study lenses are worn for a minimum of 5 days per week and 6 hours per day.

ELIGIBILITY:
Inclusion Criteria:

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

The subject must:

1. Read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Be between 18 and 39 (inclusive) years of age at the time of screening.
4. By self-report, habitually wear spherical soft silicone hydrogel contact lenses in both eyes in a daily wear or daily disposable wear modality (i.e. not extended wear modality). Habitual wear is defined as a minimum of 6 hours of wear per day, for a minimum of 5 days per week during the past 30 days.
5. Have a habitual contact lens prescription that is current within the prior 6 months, and they must have worn that prescription for at least 2 weeks prior to entering the study.
6. Possess a wearable pair of spectacles that provide correction for distance vision.

   Inclusion Criteria at Baseline Evaluation
7. The spherical equivalent of the subject's vertex-corrected distance refraction must be between -1.00 and -6.00 DS (inclusive) in each eye.
8. The magnitude of the cylindrical component of the subject's vertex-corrected distance refraction must be between 0.00 and 1.00 DC (inclusive) in each eye.
9. The best corrected, monocular, distance visual acuity must be 20/25or better in each eye.

Exclusion Criteria:

Potential subjects who meet any of the following criteria will be excluded from participating in the study: Exclusion Criteria after Screening

The subject must not:

1. Be currently pregnant or lactating.
2. Be currently using any ocular medications or have any ocular infection of any type.
3. By self-report, have any ocular or systemic disease, allergies, infection, or use of medication that the investigator believes might contraindicate or interfere with contact lens wear, or otherwise compromise study endpoints, including infectious disease (e.g., hepatitis, tuberculosis), contagious immunosuppressive disease (e.g., Human Immunodeficiency Virus [HIV]), autoimmune disease (e.g. rheumatoid arthritis, Sjögren's syndrome), or history of serious mental illness or seizures. See section 9.1 for additional details regarding excluded systemic medications.
4. Have habitually worn rigid gas permeable (RGP) lenses, orthokeratology lenses, or hybrid lenses (e.g. SynergEyes, SoftPerm) within the past 6 months.
5. Be currently wearing monovision or multifocal contact lenses.
6. Be currently wearing lenses in an extended wear modality.
7. Have participated in a contact lens or lens care product clinical trial within 30 days prior to study enrollment.
8. Be an employee (e.g., Investigator, Coordinator, Technician) or immediate family member of an employee (including partner, child, parent, grandparent, grandchild or sibling of the employee or their spouse) of the clinical site. Exclusion Criteria at Baseline Evaluation

   The subject must not:
9. Have clinically significant (grade 3 or higher on the FDA grading scale) slit lamp findings (e.g., corneal edema, neovascularization or staining, tarsal abnormalities or bulbar injection) or other corneal or ocular disease or abnormalities that the investigator believes might contraindicate contact lens wear or may otherwise compromise study endpoints (including entropion, ectropion, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, moderate or above corneal distortion, herpetic keratitis). (Specify method of determination if needed).
10. Have a history of strabismus or amblyopia.
11. Have fluctuations in vision due to clinically significant dry eye or other ocular conditions.
12. Have had or have planned (within the study period) any ocular or intraocular surgery (e.g., radial keratotomy, PRK, LASIK, iridotomy, retinal laser photocoagulation, etc.).

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 344 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (19):
- United States (19):
  - Randall Go, OD, San Francisco, California
  - Vue Optical Boutique, Jacksonville, Florida
  - Dr. James Weber & Associates, PA - City Square Blvd, Jacksonville, Florida
  - Stam & Associates Eye Care, Jacksonville, Florida
  - Sabal Eye Care, Longwood, Florida
  - Maitland Vision Center - North Orlando Ave, Maitland, Florida
  - Flora Chen Poveda, OD, PA - Orange Park, Orange Park, Florida
  - Southwest Orlando Eye Care, Orlando, Florida
  - Tallahassee Eye Center, Tallahassee, Florida
  - VisualEyes, Roswell, Georgia
  - Kannarr Eye Care, Pittsburg, Kansas
  - Birmingham Vision Care, Bloomfield, Michigan
  - Sacco Eye Group, Vestal, New York
  - ProCare Vision Centers, Granville, Ohio
  - Dr. David W. Ferris & Associates, Warwick, Rhode Island
  - Optometry Group, LLC, Memphis, Tennessee
  - Total Eye Care, Memphis, Tennessee
  - Tyler Eye Associates, Tyler, Texas
  - Botetourt Eyecare, LLC, Salem, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 344 subjects were enrolled in this study. Of those enrolled, 342 subjects were dispensed at least one study lens, while 2 subjects failed to meet all eligibility criteria. Of those dispensed, 339 subjects completed the study while 3 subjects were discontinued.
Groups:
- Test (Senofilcon A C3): Subjects randomized to receive the Test lens during the study
- Control (Delefilcon A): Subjects randomized to receive the Control lens during the study
Period: Overall Study
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
Started | 171 | 171
Completed | 169 | 170
Not Completed | 2 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Major Protocol Deviation | 1 | 0
Not completed — Subject No Longer Meets Eligibility Criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Control (Delefilcon A): Subjects that wore the Control lens during the study.
- Total: Total of all reporting groups
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A) | Total
Number analyzed (Participants) | 171 | 171 | 342
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.5 (5.44) | 30.0 (5.63) | 29.7 (5.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117 | 117 | 234
  Male | 54 | 54 | 108
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 12 | 8 | 20
  Black or African American | 15 | 15 | 30
  Native Hawaiian or Other Pacific Islander | 3 | 1 | 4
  White | 141 | 145 | 286
  Multiple | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 171 | 171 | 342

OUTCOME MEASURES:

1. Primary Outcome: End of Day Comfort
Description: End of day comfort was assessed using an individual item "Comfort at the End of the Day". Response set: Very Satisfied, Satisfied, Neither Satisfied nor Dissatisfied, Dissatisfied, and Very Dissatisfied.
Time Frame: 2-Week Follow-up
Population: All randomized subjects regardless of actual treatment and subsequent withdrawal from the study or deviation from the protocol.
Measure: Number; unit: Number of responses
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
Number analyzed (Participants) | 170 | 170
Number of responses
  Very Satisfied | 76 | 46
  Satisfied | 52 | 58
  Neither Satisfied nor Dissatisfied | 16 | 21
  Dissatisfied | 18 | 35
  Very Dissatisfied | 8 | 10
Statistical Analysis 1: Comparison: Test (Senofilcon A C3) vs Control (Delefilcon A); Test type: Superiority — Superiority was declared if the lower bound of the 2-sided 95% confidence interval is above 1; Linear Mixed Model; Odds Ratio (OR) = 2.01, 95% CI 2-sided [1.25 to 3.22] — Odds Ratio was calculated as Test over Control

2. Secondary Outcome: Digital Device Use
Description: Lens performance in digital device use was assessed using an individual item "Reduction in the feeling of tired eyes from using a computer or other digital device". Response set: Not Applicable, Excellent, Very Good, Good, Fair, and Poor. "Not Applicable" was excluded from the analysis.
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of responses
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
Number analyzed (Participants) | 170 | 170
Number of responses
  Not Applicable | 2 | 9
  Excellent | 65 | 47
  Very Good | 68 | 59
  Good | 17 | 26
  Fair | 12 | 23
  Poor | 6 | 6
Statistical Analysis 1: Comparison: Test (Senofilcon A C3) vs Control (Delefilcon A); Test type: Superiority — Superiority was declared if the lower bound of the 2-sided adjusted (96.25%) confidence interval is above 1; Linear Mixed Model; Odds Ratio (OR) = 2.00, 96.25% CI 2-sided [1.18 to 3.41] — Odds Ratio was calculated as Test over Control

3. Secondary Outcome: Comfort Throughout the Day
Description: Comfort throughout the day was measured using an individual item "I could wear these contact lenses comfortably for as long as I wanted to". Response set: Strongly Disagree, Disagree, Neither Agree Nor Disagree, Agree, and Strongly Agree.
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of responses
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
Number analyzed (Participants) | 170 | 170
Number of responses
  Strongly Disagree | 12 | 18
  Disagree | 26 | 48
  Neither Agree Nor Disagree | 16 | 17
  Agree | 43 | 43
  Strongly Agree | 73 | 44
Statistical Analysis 1: Comparison: Test (Senofilcon A C3) vs Control (Delefilcon A); Test type: Superiority — Superiority was declared if the lower bound of the 2-sided adjusted (97.5 %) confidence interval is above 1; Linear Mixed Model; Odds Ratio (OR) = 2.17, 97.5% CI 2-sided [1.30 to 3.64] — Odds Ratio was calculated as Test over Control

4. Secondary Outcome: Comfortable Vision While Night Driving
Description: Comfortable vision while night driving was assessed using an individual item "Ability to see comfortably while driving at night". Response set: Not Applicable, Excellent, Very Good, Good, Fair, and Poor. "Not Applicable" was excluded from the analysis.
Time Frame: 2-Week Follow-up
Population: as for outcome 1
Measure: Number; unit: Number of responses
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
Number analyzed (Participants) | 170 | 170
Number of responses
  Not Applicable | 2 | 3
  Excellent | 91 | 65
  Very Good | 47 | 57
  Good | 25 | 34
  Fair | 3 | 9
  Poor | 2 | 2
Statistical Analysis 1: Comparison: Test (Senofilcon A C3) vs Control (Delefilcon A); Test type: Superiority — Superiority was declared if the lower bound of the 2-sided 95% confidence interval is above 1; Linear Mixed Model; Odds Ratio (OR) = 1.77, 95% CI 2-sided [1.04 to 3.02] — Odds Ratio was calculated as Test over Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; The study duration for each subject was approximately 2 weeks.
Arm/Group | Test (Senofilcon A C3) | Control (Delefilcon A)
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/171
Serious Adverse Events (participants affected / at risk) | 0/171 | 0/171
Other Adverse Events (participants affected / at risk) | 0/171 | 0/171

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT05300763/Prot_SAP_000.pdf